CLINICAL TRIAL: NCT01607502
Title: Database for Clinical and Anamnestic Data in Pulmonary Hypertension
Status: Recruiting | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: 23-408 ex 10/11
Record Dates: First submitted 2012-04-13; First posted 2012-05-30 (Estimated); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Pulmonary Hypertension
Keywords: Pulmonary hypertension; database; biomarker
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples are collected and stored anonymously in our biobank if patients give their informed consent containing the option of DNA analysis.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients of our outpatient clinic: Patients who have an investigation in our outpatient clinic for pulmonary hypertension like a echocardiography, a right heart catheterization or a cardio pulmonary exercise testing

SUMMARY:
Pulmonary hypertension (PH) is defined as a pulmonary arterial mean pressure (meanPAP) ≥ 25 mmHg measured in the right heart catheterization.

There are different forms of PH defined in the classification of Dana Point 2008.

PH is diagnosed with right heart catheterization but there are other non invasive methods which can be used for screening like the echocardiography, stress echocardiography and cardio pulmonary exercise testing. In the diagnosis process and in the follow up of PH patients biomarkers like NTproBNP are helpful. There are no specific biomarkers for the disease which can make the diagnosis process easier and predict prognosis.

The systematic data collection in a data base provides better information about patients in daily routine and clinical studies as well as in the design of new studies.

DETAILED DESCRIPTION:
In this study the investigators want to collect clinical data of PH patients and controls in a database as well as blood samples in a biobank. The combination of anamnestic and clinical data and biomarkers should provide a better characterization of our patients and should improve the analysis of the disease development of different PH forms and therapeutic aspects.

After given informed consent patients' data are entered in a database at different time points. The database includes parameter of several invasive and non-invasive investigations like right heart catheterization (RHC), echocardiography, ECG, pulmonary function tests, cardiorespiratory exercise testing, 6-minute walk test, computed tomography, MRI, polysomnography, blood gas analysis and laboratory data as well as demographic data of the patients.

The blood samples are taken during routine punctuation and are stored in our biobank.

ELIGIBILITY:
Inclusion Criteria:

* patients with pulmonary hypertension
* patients at risk for getting pulmonary hypertension
* patients who have symptoms which my be due to pulmonary hypertension when we have their written informed consent.

Exclusion Criteria:

* patients without written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who come to our outpatient clinic with pulmonary haypertension, symptoms that may be caused by pulmonary hypertension and patients at risk for pulmonary hypertension
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2010-07; Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Collecting data in a PH patient database | After one year: first analysis of retrospectively collected data. Ongoing data collection: new data of patients who are already in the database, new patients (3-4 years)
  Retrospective and prospective data input and constant update

CONTACTS AND LOCATIONS:
Overall Officials: Horst Olschewski, MD, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University of Graz, Graz, Austria

REFERENCES:
- [Derived] Kovacs G, Avian A, Foris V, Tscherner M, Kqiku X, Douschan P, Bachmaier G, Olschewski A, Matucci-Cerinic M, Olschewski H. Use of ECG and Other Simple Non-Invasive Tools to Assess Pulmonary Hypertension. PLoS One. 2016 Dec 28;11(12):e0168706. doi: 10.1371/journal.pone.0168706. eCollection 2016. PMID 28030578